CLINICAL TRIAL: NCT01344681
Title: A Randomized Phase II, Multi-center, Non-inferiority Clinical Trial for Efficacy and Safety of Micafungin Versus Intravenous Itraconazole as Empirical Antifungal Therapy for Febrile Neutropenic Patients With Hematological Diseases
Brief Title: Micafungin Versus Intravenous Itraconazole as Empirical Antifungal Therapy for Febrile Neutropenic Patients With Hematological Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0794
Record Dates: First submitted 2011-04-25; First posted 2011-04-29 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Febrile Neutropenia; Hematological Diseases
MeSH Terms: conditions — Febrile Neutropenia; Hematologic Diseases | interventions — Micafungin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Micafungin sodium
  Interventions: Drug: Micafungin sodium
- Arm B (Active Comparator): Itraconazole
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Micafungin sodium — 1. Treatment period (active treatment): an average 14 days
  2. Dosage:
     - Study Drug: Micafungin sodium (mycamine ® injections 50mg/vial) 2 vials (100mg / day)
  3. Administration Method:
     * Study Drug: 3-5 days after fever begins. Infusion one time a day (one hour). Termination of treatment after maintaining fever for three days or the recovery of neutrophils with no fever.
  Other Names: Mycamine®
  Arms: Arm A
Drug: Itraconazole — 1. Treatment period (active treatment): an average 14 days
  2. Dosage:
     - Active Comparator: Itraconazole (Sporanox ® injection) 200 mg 2 times(400mg / day)
  3. Administration Method:
     * Active Comparator: 200 mg two times(400 mg) a day, total of 4 times for 2 days and then one times (200 mg) a day for 12 days. Termination of treatment after keeping fever for three days or the recovery of neutrophils with no fever.
  Other Names: Sporanox®
  Arms: Arm B

SUMMARY:
This study of chemotherapy occurred during the neutropenic fever in patients with antibiotic refractory fever. The investigators evaluate efficacy and safety of micafungin sodium (mycamine ® Injection) 100mg dose compare to itraconazole (Sporanox ® Injection) 200mg as a control and this study is prospective, randomized, non-inferiority trials.

Therefore, this study was planned for review of the safety and efficacy in korean patients.

ELIGIBILITY:
Inclusion Criteria:

* The male and female patients over 18 years
* To participate in clinical trials and voluntary written consent requirement to comply with a patient
* Chemotherapy with a variety of hematologic malignancies or patients undergoing stem cell transplantation
* Fever (temperature ≥ 38.4 ℃) showing Neutropenia (absolute neutrophil count <500/mm3) patients
* Combined antibiotic therapy 72 hours after the expiration of term lasts three patients

Exclusion Criteria:

* Of clinical trials of breast-feeding or pregnant women of childbearing age with intent to
* Adapted species (candida genus, aspergillus genus) Colitis caused by fungi other than the patients with fungal infection
* HIV-positive patient serum
* This test within 30 days of assignment to the other patients participating in clinical trials
* Within 72 hours of registration before the patients treated with systemic antifungal agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Responses to therapy | 7 days after stopping study medication
  1. definition of 'treatment success': (5 Items to meet all your success)
     * Within 7 days after stopping study medication if there is no fungal infection
     * 7 days after stopping study medication if you are alive
     * Neutropenia period of serious adverse events or lack of effective medication is not stopped
     * If fever during neutropenia (temperature <37.5 ℃)
     * Treatment until the end of the existing fungal infection is treated completely or partially
  2. definition of 'treatment failure': - If you failed any of 5 Items in 'treatment success'

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Dong-A Medical Center, Busan
  - Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - ASAN Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Medical Center, Suwon